CLINICAL TRIAL: NCT04022993
Title: An Open-label, Randomized, Multi-center, Parallel-group Clinical Trial Comparing the Efficacy and Safety of Insulin RinGlar® ("Geropharm", Russia) Compared to Lantus® SoloStar® ("Sanofi-Aventis Deutschland GmbH", Germany) in Type 1 Diabetes Mellitus Patients
Brief Title: Efficacy and Safety of Insulin RinGlar® Compared to Lantus® SoloStar® in Type 1 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLARGIN-IM
Record Dates: First submitted 2019-07-05; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-01

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus
Keywords: Diabetes Mellitus, Type 1; Insulin; Glargine
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lantus® SoloStar® (Active Comparator): Lantus® SoloStar® once a day, individually glucose-level based administered in stable doses, started before enrollement
  Interventions: Drug: Lantus Solostar, 100 Units/mL Subcutaneous Solution
- Insulin RinGlar® (Experimental): Insulin RinGlar® once a day, individually glucose-level based administered in stable doses, started before enrollement
  Interventions: Drug: Insulin RinGlar, 100 Units/mL Subcutaneous Solution

INTERVENTIONS:
Drug: Lantus Solostar, 100 Units/mL Subcutaneous Solution — 4 weeks of glucose-level based dose titration, 22 weeks of treatment with stable doses
  Arms: Lantus® SoloStar®
Drug: Insulin RinGlar, 100 Units/mL Subcutaneous Solution — 4 weeks of glucose-level based dose titration, 22 weeks of treatment with stable doses
  Arms: Insulin RinGlar®

SUMMARY:
The study is designed to approve non-inferior efficacy and safety of Insulin RinGlar® compared to Lantus® SoloStar® in Type 1 Diabetes Mellitus Patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed written consent
* Diabetes mellitus type 1 for at least 12 months prior to screening
* History of basis-bolus (multiple dose injection (MDI)) therapy in stable doses at least 30 days
* Glycated hemoglobin (HbA1c) level of 6.5 to 12.0 % at screening (both values inclusive)
* Body mass index (BMI) of 18.0 to 35 kg/m2 at screening (both values inclusive)
* Subject is able and willing to comply with the requirements of the study protocol

Exclusion Criteria:

* Contraindication to the use of Insulin glargine
* Insulin resistance over 1.5 U/kg insulin pro day
* History of treatment any biosimilar insulin
* History of treatment any experimental drugs or medical devices for 3 months prior to screening
* History of treatment insulin pump for 90 days prior to signed written consent or indication for use insulin pump
* Presence of severe diabetes complications
* History of severe hypoglycemia during 6 months prior to signed written consent
* History of 15 or more episodes mild hypoglycemia during 1 month prior to signed written consent
* History or presence of uncontrolled diabetes mellitus for 6 months prior to screening
* History of administration of glucocorticoids for 1 year prior to screening
* Administration of any immunosupressive drugs (Cyclosporinum, Methotrexatum, etc.)
* History of autoimmune disease, except vitiligo and controlled autoimmune polyglandular syndrome (APS) types 1-3, except adrenal insufficiency
* History of hypersensitivity to any of the active or inactive ingredients of the insulin/insulin analogue preparations used in the trial, OR history of significant allergic drug reactions
* History of severe allergic reactions
* Pregnant and breast-feeding women
* Acute inflammation disease for 3 weeks prior to screening
* Deviation of the laboratory results conducted during the screening:

Hemoglobin value < 9,0 g/dl; Hematocrit value < 30 %; ALT and AST value > 2 folds as high as maximal normal value; Serum bilirubin value > 1.5 folds as high as maximal normal value

* History of hematological disorders that can affect the reliability of HbA1c estimation (hemoglobinopathies, hemolytic anemia, etc.)
* Serious blood loss for 3 months prior to screening (blood donation, surgery procedure, etc.)
* Incomplete recovery after surgery procedure
* History of unstable angina, myocardial infarction, severe arrhythmia, heart failure III or IV NYHA for 1 year prior to screening
* History of stroke or TIA for 6 months prior to screening
* History of drug, alcohol abuse for 3 years prior to screening
* Inability follow to protocol
* History of oncological disease during 5 years prior to screening
* Serological evidence of human immunodeficiency virus (HIV), hepatitis B (HbSAg), hepatitis C (HCVAb) or syphilis (Treponema pallidum) antibodies at screening.
* History of transplantation, except 3 months after corneal transplant
* History or presence of a medical condition or disease that in the investigator's opinion would embarrass glycemic control and completion of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Antibody Response | 26 weeks
  Change from baseline in titer of antibodies to human insulin

SECONDARY OUTCOMES:
Adverse Events frequency and degree | 26 weeks (4+22 weeks)
  Hypoglycemic episodes (glucose level < 3.9 mmol/l) frequency; Occurrence of local reactions at injection sites; Occurrence allergic reactions.
Glycated hemoglobin | 26 weeks
  Change in HbA1c from baseline
Fasting Plasma Glucose Level | 26 weeks
  Change in fasting plasma glucose level from baseline
Seven-Point Glucose Testing | 26 weeks
  Change in seven-point glucose testing results from baseline
Basal Insulin Dose | 26 weeks
  Change in basal insulin dose per body weight (U/kg) from baseline
Total Insulin Dose | 26 weeks
  Change in total insulin dose per body weight (U/kg) from baseline
Body Mass Index | 26 weeks
  Change in BMI from baseline
Treatment Satisfaction | 26 weeks
  Change in overall treatment satisfaction (DTSQ score) from baseline
Achievement of Glycated Hemoglobin Goals | 26 weeks
  The frequency of achievement glycated hemoglobin goals
Achievement of Glycated Hemoglobin < 7% | 26 weeks
  The frequency of achievement glycated hemoglobin < 7% ( 7% inclusive)

CONTACTS AND LOCATIONS:
Overall Officials: Tatyana L Karonova, MD, DSc, Principal Investigator — Almazov National Medical Research Centre
Locations (14):
- Russia (14):
  - Arkhangelsk Regional Clinical Hospital, Arkhangelsk
  - Kazan Endocrinology Dispensary, Kazan'
  - Krasnoyarsk State Medical University named after Professor V.F. Voino-Yasenetsky, Krasnoyarsk
  - Endocrinology Research Centre (Moscow), Moscow
  - V.A. Baranov Republic Hospital, Petrozavodsk
  - Rostov State Medical University, Rostov-on-Don
  - Polyclinic Сomplex, Saint Petersburg
  - City Diagnostic Center № 1, Saint Petersburg
  - City Hospital № 2, Saint Petersburg
  - City Polyclinic № 117, Saint Petersburg
  - EosMed, Saint Petersburg
  - Almazov National Medical Research Centre, Saint Petersburg
  - Pokrovskaya Municipal Hospital, Saint Petersburg
  - Clinical City Hospital № 9, Saratov

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karonova TL, Mosikian AA, Mayorov AY, Makarenko IE, Zyangirova ST, Afonkina OA, Belikova TM, Zalevskaya AG, Khokhlov AL, Drai RV. Safety and efficacy of GP40061 compared with originator insulin glargine (Lantus(R)): a randomized open-label clinical trial. J Comp Eff Res. 2020 Mar;9(4):263-273. doi: 10.2217/cer-2019-0136. Epub 2020 Feb 6. PMID 32027167